CLINICAL TRIAL: NCT01621971
Title: Comparative Effects of Brief Inhaled Milrinone Versus Intravenous Milrinone on Pulmonary Arterial Pressure in Patients Undergoing Mitral Valve Surgery
Brief Title: Effect of Brief Nebulization of Milrinone on Pulmonary Arterial Pressure Before Cardiopulmonary Bypass on Mitral Valve Surgery Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH-MI201106
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Hypertension; Mitral Regurgitation
Keywords: inhaled milrinone; pulmonary hypertension; mitral regurgitation; mitral valve surgery
MeSH Terms: conditions — Hypertension, Pulmonary; Mitral Valve Insufficiency | interventions — Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- milrinone inhalation (Experimental): inhaled milirinone and IV placebo (0.9% normal saline 0.05 ml/kg) are administered in Group IH.
  Interventions: Drug: inhaled milrinone
- intravenous milrinone (Active Comparator): After performing the sternotomy and achieving stable hemodynamics, but before the initiation of CPB, inhaled placebo (distilled water) and an IV bolus of milrinone (50 μg/kg) are administered in Group IV
  Interventions: Drug: intravenous milrinone

INTERVENTIONS:
Drug: inhaled milrinone — After performing the sternotomy and achieving stable hemodynamics, but before the initiation of CPB, inhaled milirinone and intravenous placebo (0.9% normal saline 0.05 ml/kg) are administered
  Other Names: Primacor, Sanofi-Synthelabo Canada Inc., Markham, ON, Canada
  Arms: milrinone inhalation
Drug: intravenous milrinone — After performing the sternotomy and achieving stable hemodynamics, but before the initiation of CPB, inhaled placebo (distilled water) and an intravenous bolus of milrinone (50 μg/kg) are administered
  Other Names: Primacor, Sanofi-Synthelabo Canada Inc., Markham, ON, Canada
  Arms: intravenous milrinone

SUMMARY:
Our main hypothesis is that inhalation of milrinone can reduce the elevated pulmonary arterial pressure due to severe mitral valve regurgitation without compromising systemic hemodynamics. Therefore, the effects of a brief inhaled milrinone (IH) on pulmonary artery pressure are determined and compared to those of intravenous milrinone (IV) in severe mitral regurgitation patients undergoing mitral valve surgery.

DETAILED DESCRIPTION:
Perioperative pulmonary hypertension (PHT), an independent risk factor for cardiac surgery, 1,2 is frequently associated with chronic mitral valve regurgitation and tends to produce right ventricular (RV) dysfunction. Worsening PHT, which is sensitive to any increase in the RV afterload, reduces the right coronary perfusion pressure, exacerbates RV dysfunction, and compromise the left ventricular (LV) preload and systemic perfusion pressure. 3,4 Although intravenous (IV) milrinone is preferred for treating PHT due to its beneficial effects in enhancing myocardial contractability without increasing the heart rate-related myocardial oxygen consumption, 5-7 its frequent association with systemic vasodilation requires additional vasoconstrictor therapy for maintaining the optimal perfusion pressure.8-10 Selective pulmonary vasodilation, which reduces the RV afterload without systemic arterial vasodilation, is important for managing PHT and the accompanying RV dysfunction.11 A study reported that nebulized and inhaled (IH) milrinone ( 1 mg/ml) produced dose-dependent selective pulmonary vasodilatation in postoperative PHT in the intensive care unit.12 If IH milrinone during the pre-cardiopulmonary bypass (CPB) period produces selective pulmonary vasodilation in patients with PHT undergoing mitral valve surgery, it would be a beneficial option for managing intraoperative PHT.

Our main hypothesis is that a brief inhaled milrinone could reduce the pulmonary arterial pressure without the systemic side effects better than intravenous milrinone in elevated pulmonary artery pressure patients. The aim of this study is to determine the effects of hemodynamic before and after administering IH and to compare them to those of IV milrinone in patients with elevated pulmonary artery pressure due to severe mitral regurgitation undergoing mitral valve surgery.

Materials and Methods Experimental Groups Adult patients with PHT (systolic PAP > 50 mmHg estimated by the velocity of tricuspid valve regurgitation in preoperative transthoracic echocardiography) undergoing mitral valve surgery for chronic mitral regurgitation are enrolled in this study after obtaining approval from the institutional research board and providing written informed consent.

Preoperative exclusion criteria include preoperative supraventricular tachycardia (SVT), atrial fibrillation, atrial flutter, multiple ventricular ectopic contractions, continuous inotropic support, LV ejection fraction (EF) < 30%, emergent surgery, obstructive cardiomyopathy, bleeding diatheses, bronchial asthma and had biochemical evidence of hepatic disease or renal impairment.

The pharmacist implements the randomization process for grouping the patients by giving the enrolled patients, a patient identification number (PIN). Then, the patients are stratified by their PIN in a 1:1 ratio to receive IH (Primacor, Sanofi-Synthelabo Canada Inc., Markham, ON, Canada) (Group IH) or IV (Group IV) milrinone. The investigators are blinded to the allocation of the study group.

Anesthesia and Patient Monitoring When the patient arrived in the operating room, continuous monitoring of a five-lead ECG (lead II and V5), the bispectral index (BIS), pulse oximetry, and invasive arterial pressure via the radial artery are started. Patients are given midazolam 1.5-2 mg intravenously in the patient holding area. Anesthesia is induced with propofol 1-1.5 mg/kg, fentanyl 10-15 μg/kg, and rocuronium 0.9 mg/kg. Target controlled infusion (TCI) and a TCI infusor (Diprifusor™ TCI system; Fresenius, Waltham, MA, USA) are used to administer propofol for anesthetic induction and maintenance, and the infusion dose is titrated to achieve a propofol effect-site concentration of 2-2.5 μg/ml. Additional fentanyl at 10-30 μg/kg/h and rocuronium at 20-30 mg/h are administered to maintain anesthesia, and the propofol concentration is adjusted to maintain a BIS score of 40-60. After tracheal intubation, volume-controlled ventilation of oxygen with air (FiO2 0.6, flow rate 100 ml/kg/min) is started with a tidal volume of 10 ml/kg, respiration rate of 12-14/min, inspiration:expiration ratio of 1:2, and peak airway pressure lower than 25 cmH2O. Then, the respiration rate is adjusted to maintain an end-tidal CO2 of 35-40 mmHg.

An introducer and a pulmonary artery catheter (Oximetrix™ Opticath catheter; Abbot Laboratories, North Chicago, IL, USA) are placed in the right internal jugular vein. A transesophageal echocardiography (TEE) probe is placed, and intraoperative TEE is used to monitor ventricular and valvular function throughout the operation. The LV EF is measured using a modification of Simpson's method from the midesophageal 4 or 2 chamber view of two-dimensional TEE images as appropriate.

During and after anesthesia induction and obtaining vascular access for hemodynamic monitoring, synthetic hydroxyethylstarch (Voluven™; Fresenius Kabi, Bad Homberg, Germany) is administered as needed to maintain stable hemodynamics, and bolus phenylephrine 50-100 μg is administered intravenously to treat any refractory hypotension (MAP < 60 mmHg) persisting for more than 1 min with intravascular volume administration.

After delivering the study drugs and collecting data, CPB with moderate hypothermia (rectal temperature 28-30ºC) via crystalloid cardioplegia is used during the surgical procedure. The MAP was maintained at 50-80 mmHg by adjusting the pump flow and administering 50 μg boluses of phenylephrine during the CPB period.

The IV milrinone infusion (0.5 μg/kg/min) is started at the release of the aortic cross-clamp and a continuous infusion of norepinephrine is started at a rectal temperature of 35ºC as needed; its dosage is titrated to wean the patient from CPB and to maintain the optimal hemodynamics during the post-CPB period in both groups.

Delivery of the Study Drug After performing the sternotomy and achieving stable hemodynamics, but before the initiation of CPB, the study drugs are administered; IH milirinone and IV placebo (0.9% normal saline 0.05 ml/kg) or IH placebo (distilled water) and an IV bolus of milrinone (50 μg/kg) are administered in Group IH and IV, respectively. Milrinone is used at its commercial concentration (1.0 mg/ml) for both inhalation and IV administration. The reservoir of a nebulizer (MiniHeart™; Westmed, Tucson, AZ, USA) in the inspiratory limb of the ventilator circuit (90 cm proximal to the Y-piece) is filled with milrinone or placebo. The milrinone or placebo in the reservoir is nebulized with a fixed operating flow at 2 L/min of O2 (as per the manufacturer's recommendation) and delivered over 10 min at a ventilator flow rate of 100 ml/kg/min to avoid rebreathing the expiratory flow, which may produce contamination or interaction between the nebulized milrinone and CO2 absorbent (Fig. 1). The aerosol size and delivery rate of the nebulized drug are assumed to be 1.0-2.5 μm and 45-65 μL per gas flow, respectively, according to the manufacturer's manual for the nebulizer. Excess inspiratory gas flow from the nebulizer was compensated for by adjustment of minute ventilation settings on the ventilator, keeping minute ventilation constant. Inspiratory oxygen fraction (FiO2) is kept constant throughout the procedure. If MAP decreases below 60 mmHg, inhalation of the study drug is stopped and the patient excluded from the study.

Hemodynamic Data The following data are obtained before and 10 min after completely administering the study drug: mean arterial pressure (MAP), mean pulmonary arterial pressure (MPAP), central venous pressure (CVP), pulmonary arterial occlusion pressure (PAOP), the transpulmonary pressure gradient (TPG= mean PAP-PAOP), thermodilution cardiac output (CO), systemic vascular resistance (SVR), pulmonary vascular resistance (PVR), arterial O2 tension (PaO2), mixed venous O2 saturation (SvO2), and TEE measured EF.

Statistical Analysis Intergroup comparisons of the changes in SVR, PVR, the PVR/SVR ratio, and TPG are used to identify selective pulmonary vasodilation. The data before and after administration are compared using paired t-test. If the data do not pass a normality test, the Wilcoxon signed-rank test was used. Intergroup data are compared using the t-test. The need for bolus phenylephrine due to hypotension in the pre-CPB period or during CPB is compared using Fisher's exact test. Statistical significance is assumed at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing mitral valve surgery for chronic mitral regurgitation
* estimated pulmonary hypertension (systolic PAP > 50 mmHg estimated by the velocity of tricuspid valve regurgitation in preoperative transthoracic echocardiography)
* patients who agreed to participate in this study and signed written informed consent

Exclusion Criteria:

* preoperative supraventricular tachycardia (SVT),
* atrial fibrillation,
* atrial flutter,
* multiple ventricular ectopic contractions,
* continuous inotropic support,
* LV ejection fraction (EF) < 30%,
* emergent surgery,
* obstructive cardiomyopathy,
* bronchial asthma
* biochemical evidence of hepatic disease or renal impairment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
transpulmonary pressure gradient | 10 min after milrinone administration
  transpulmonary pressure gradient (TPG= mean PAP-PAOP) before and 10 min after completely administering the study drug

SECONDARY OUTCOMES:
mean pulmonary arterial pressure | 10 min after milrinone administration
  mean pulmonary artery pressure (MPAP) before and 10 min after completely administering the study drug
mean arterial pressure | 10 min after milrinone administration
  mean arterial pressure(MAP) before and 10 min after completely administering the study drug
systemic vascular resistance | 10 min after milrinone administration
  systemic vascular resistance (SVR) before and 10 min after completely administering the study drug
pulmonary vascular resistance | 10 min after milrinone administration
  pulmonary vascular resistance (PVR) before and 10 min after completely administering the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea